CLINICAL TRIAL: NCT04262050
Title: The Effect of Combination Transcranial Direct Current Stimulation and Transcranial Magnetic Stimulation on Subjective Tinnitus and Combined Depression
Brief Title: Combined tDCS and TMS on Subjective Tinnitus and Combined Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Jin Song, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1607/355-004
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Tinnitus; Depression
Keywords: Tinnitus, tDCS, TMS
MeSH Terms: conditions — Tinnitus; Depression | interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (4):
- TMS + tDCS group (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS)
- sham TMS + tDCS group (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS)
- tDCS group (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS)
- TMS group (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS)

SUMMARY:
The investigators combined transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS) to increase the effective response of a single session of neuromodulation in subjective tinnitus.

DETAILED DESCRIPTION:
To treat motor and psychiatric disorders, transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS) are world-widely in use in clinics. The investigators combined these two types of neuromodulation techniques to increase the effective response of a single session of neuromodulation in subjective tinnitus. Experimental groups with 80 tinnitus subjects consisted of four different treatment groups which are tDCS, tDCS with sham TMS, tDCS-TMS and TMS group. Subjects were given 1.5milliampere (mA) tDCS on the bi-frontal area and TMS stimulated contralateral single side of the temporoparietal cortex with 200 pulses at 1herz (Hz) stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Research volunteers who agreed to participate in the clinical trial were gathered from the tinnitus clinic of the Department of Otorhinolaryngology Head-and-Neck Surgery, Seoul National University Bundang Hospital

Exclusion Criteria:

* psychoactive drug user
* implanted material
* pacemaker user

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Tinnitus handicap inventory | the same 1 day after treatment
  tinnitus-related questionnaire

IPD SHARING:
Plan to Share IPD: No